CLINICAL TRIAL: NCT01490866
Title: A Phase II Trial of Single Agent Axitinib as Maintenance Therapy for Patients With First Line Metastatic Colorectal Cancer (mCRC)
Brief Title: A Trial of Single Agent Axitinib as Maintenance Therapy for Patients With First Line Metastatic Colorectal Cancer (mCRC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GI 154
Record Dates: First submitted 2011-11-07; First posted 2011-12-13 (Estimated); Results first posted 2017-01-12 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; Axitinib; FOLFOX/Bevacizumab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Axitinib; Bevacizumab; Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FOLFOX/bevacizumab and Axitinib (Experimental): Phase II trial investigating axitinib as a single-agent maintenance therapy following standard first-line FOLFOX/bevacizumab therapy for patients with mCRC. (FOLFOX is a combination of 5-Fluorouracil, Leucovorin and Oxaliplatin.)
  All patients will receive FOLFOX/bevacizumab for four 28-day cycles (a total of 16 weeks). After 4 cycles, maintenance axitinib will be started.
  Interventions: Drug: Axitinib; Drug: Bevacizumab; Drug: 5-Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Axitinib — 5-mg tablets PO BID
  Other Names: AG-013736
Drug: Bevacizumab — 5 mg/kg Days 1 and 15; IV
  Other Names: Avastin
Drug: 5-Fluorouracil — 400 mg/m2 Days 1 and 15; IV
  Other Names: 5-FU
Drug: 5-Fluorouracil — 2400 mg/m2 over 46-48 hours Days 1 and 15; Continuous Intravenous
  Other Names: 5-FU
Drug: Leucovorin — 400 mg/m2 Days 1 and 15; IV
  Other Names: folinic acid
Drug: Oxaliplatin — 85 mg/m2 Days 1 and 15; IV
  Other Names: Eloxatin

SUMMARY:
This is a non-randomized, open-label, Phase II trial investigating axitinib as a single-agent maintenance therapy following standard first-line FOLFOX/bevacizumab therapy for patients with mCRC.

DETAILED DESCRIPTION:
All patients will receive FOLFOX/bevacizumab for four 28-day cycles (a total of 16 weeks). After 4 cycles, maintenance axitinib will be started. With approval of the Medical Monitor,patients who are having significant benefit from FOLFOX/bevacizumab may continue chemotherapy to a maximum of six 28-day cycles. During trial treatment, all patients will be assessed for response every 8 weeks (2 cycles).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic adenocarcinoma of the colon or rectum.
* Patients must have measurable disease per RECIST Version 1.1.
* No previous systemic therapy for metastatic colorectal cancer. Previous radiosensitizing chemotherapy is allowed, if completed at least 4 weeks prior to Cycle 1 Day 1 of study treatment, and previous neoadjuvant and/or adjuvant chemotherapy is allowed, if completed at least 6 months prior to diagnosis of metastatic disease.
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 to 1.
* Life expectancy >=12 weeks.
* Adequate hematologic, renal and hepatic function
* Patients who are on coumadin should have an INR value within the therapeutic range (i.e., 2 to 3 x ULN). Patients who are on stable, chronic doses of coumadin are eligible.
* Male patients willing to use adequate contraceptive measures. Female patients who are not of child-bearing potential, and female patients of child-bearing potential who agree to use adequate contraceptive measures, who are not breastfeeding, and who have a negative serum or urine pregnancy test performed within 72 hours prior to start of treatment.
* Willingness and ability to comply with the trial and follow-up procedures.
* Ability to understand the investigative nature of this trial and give written informed consent.

Exclusion Criteria:

* History or known presence of central nervous system (CNS) metastases.
* Patients who have had a major surgical procedure (not including mediastinoscopy), or significant traumatic injury <=4 weeks prior to beginning treatment.
* Women who are pregnant or lactating. All females of child-bearing potential must have negative serum or urine pregnancy tests within 72 hours prior to study treatment (see Appendix D)
* History of hypersensitivity to active or inactive excipients of any component of treatment (5 fluorouracil, bevacizumab, oxaliplatin, or axitinib), or known dipyrimidine dehydrogenase deficiency.
* Patients with proteinuria at screening as demonstrated by:

  * Urine dipstick for proteinuria >=2+ (patients discovered to have >=2+ proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection, and must demonstrate <=1 g of protein/24 hours to be eligible)
* Patients with a serious non healing wound, active ulcer, or untreated bone fracture.
* Patients with evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation).
* Patients with history of hematemesis or hemoptysis (defined as having bright red blood of ½ teaspoon or more per episode) <=1 month prior to study enrollment.
* Patients requiring concomitant treatment with potent CYP3A4 or CYP1A2 inducers and CYP3A4 inhibitors.
* History of myocardial infarction or unstable angina <=6 months prior to beginning treatment.
* Inadequately controlled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg while on antihypertensive medications). Initiation of antihypertensive agents is permitted provided adequate control is documented at least 1 week prior to Day 1 of study treatment.
* New York Heart Association Grade II or greater congestive heart failure.
* Serious cardiac arrhythmia requiring medication. Patients with chronic, rate-controlled atrial fibrillation are eligible.
* Significant vascular disease (e.g., aortic aneurysm requiring surgical repair, or recent peripheral arterial thrombosis) <=6 months prior to Day 1 of treatment.
* History of stroke or transient ischemic attack <=6 months prior to beginning treatment.
* Any prior history of hypertensive crisis or hypertensive encephalopathy.
* History of abdominal fistula or gastrointestinal perforation <=6 months prior to Day 1 of beginning treatment.
* Concurrent severe, intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.
* Any known positive test for human immunodeficiency virus, hepatitis C virus or acute or chronic hepatitis B infection.
* Mental condition that would prevent patient comprehension of the nature of, and risk associated with, the study.
* Use of any non-approved or investigational agent <=28 days prior to administration of the first dose of study drug. Patients may not receive any other investigational or anti-cancer treatments while participating in this study.
* Past or current history of neoplasm other than the entry diagnosis with the exception of treated non-melanoma skin cancer or carcinoma in situ of the cervix, or other cancers cured by local therapy alone and a disease free survival >=5 years.
* Infection requiring IV antibiotics.
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter drug absorption (e.g. active inflammatory bowel disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or significant small bowel resection).
* Inability to swallow whole tablets.
* Patients with > Grade 2 peripheral neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Bendell, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (12):
- United States (12):
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - Florida Cancer Specialists-South, Fort Myers, Florida
  - Woodlands Medical Specialists, Pensacola, Florida
  - Florida Cancer Specialists-North, St. Petersburg, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Oncology Hematology of SW Indiana, Newburgh, Indiana
  - Hope Cancer Center, Terre Haute, Indiana
  - Grand Rapids Oncology Program, Grand Rapids, Michigan
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Atlantic Health System, Summit, New Jersey
  - Tennessee Oncology, Nashville, Tennessee
  - Texas Health Physician Group, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between January 2012 and January 2014, 70 patients with histologically or cytologically confirmed metastatic carcinoma of colon or rectum were enrolled and treated. The trial was conducted at 12 sites in the United States.
Pre-assignment Details: In this non-randomized open label trial, patients began treatment with FOLFOX/bevacizumab every 4 weeks for 16 weeks. Patients with objective response or stable disease began Axitinib maintenance therapy at week 17. Axitinib therapy continued until disease progression, unacceptable toxicity or did not meet any criteria for discontinuation.
Groups:
- FOLFOX/Bevacizumab and Axitinib: All patients receive FOLFOX/bevacizumab for four 28-day cycles (16 weeks). After 4 cycles, axitinib maintenance will be administered starting on Week 17. Maintenance treatment will continue until disease progression or intolerable toxicity occurs.
  FOLFOX/bevacizumab ( FOLFOX is a combination of Leucovorin, fluorouracil and oxiloplatin):
  * 5-Fluorouracil: 400 mg/m2 Days 1 and 15 by IV followed by 2400 mg/m2 over 46-48 hours Days 1 and 15 by continuous infusion;
  * Leucovorin: 400 mg/m2 given Days 1 and 15 by IV
  * Oxaliplatin: 85 mg/m2 Days 1 and 15 by IV
  * Bevacizumab: 5 mg/kg on Days 1 and 15 by IV
  Maintenance:
  - Axitinib: 5-mg tablets orally twice per day on Days 1 thru 28 of each cycle until disease progression or unacceptable toxicity occurs.
Period: FOLFOX/Bevacizumab Treatment
Arm/Group | FOLFOX/Bevacizumab and Axitinib
Started | 70
Completed | 49
Not Completed | 21
Not completed — Disease Progression | 6
Not completed — Adverse Event | 6
Not completed — Withdrawal by Subject | 5
Not completed — Protocol Violation | 1
Not completed — Intercurrent illness | 1
Not completed — Physician Decision | 2
Period: Axitinib Maintenance Therapy
Arm/Group | FOLFOX/Bevacizumab and Axitinib
Started | 49
Completed | 0 (No protocol defined endpoint to Axitinib maintenance treatment.)
Not Completed | 49
Not completed — Disease Progression | 30
Not completed — Adverse Event | 12
Not completed — Withdrawal by Subject | 3
Not completed — Protocol Violation | 2
Not completed — Intercurrent illness | 2

BASELINE CHARACTERISTICS:
Groups:
- FOLFOX/Bevacizumab and Axitinib: All patients receive FOLFOX/bevacizumab for four 28-day cycles (a total of 16 weeks). After 4 cycles, axitinib maintenance will be administered. FOLFOX is a combination of Leucovorin, fluorouracil and oxiloplatin.
  FOLFOX/bevacizumab:
  * 5-Fluorouracil: 400 mg/m2 Days 1 and 15 by IV followed by 2400 mg/m2 over 46-48 hours Days 1 and 15 by continuous infusion;
  * Leucovorin: 400 mg/m2 given Days 1 and 15 by IV
  * Oxaliplatin: 85 mg/m2 Days 1 and 15 by IV
  * Bevacizumab: 5 mg/kg on Days 1 and 15 by;IV
  Maintenance:
  - Axitinib: 5-mg tablets orally twice per day (PO BID)
Arm/Group | FOLFOX/Bevacizumab and Axitinib
Number analyzed (Participants) | 70
Age, Continuous [Median (Full Range); unit: years] | 60 [36 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 36
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 62
  Black/African American | 6
  Asian | 1
  Unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Defined as the time from first treatment until objective tumor progression or death from any cause, assessed according to Response Evaluation Criteria for Solid Tumors (RECIST) v1.1.
Time Frame: 24 months
Population: All patients who received at least one dose of any study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FOLFOX/Bevacizumab and Axitinib
Number analyzed (Participants) | 70
months | 8.3 [7.8 to 9.4]

2. Secondary Outcome: Objective Response Rate
Description: Defined as the percentage of evaluable patients showing a complete or partial response (CR or PR) per RECIST v1.1 criteria. CR = disappearance of all lesions. PR = at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Stable disease (SD) = neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest (nadir) sum LD since start of treatment.
Time Frame: every 8 weeks, assessed up to approximately 24 months
Measure: Number; unit: percentage of participants
Arm/Group | FOLFOX/Bevacizumab and Axitinib
Number analyzed (Participants) | 61
percentage of participants
  Objective Response | 34
  Stable Disease | 57

3. Secondary Outcome: Time To Progression (TTP)
Description: Defined as the time after a disease is diagnosed (or treated) until worsening of the disease.
Time Frame: every 8 weeks, assessed approximately up to 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FOLFOX/Bevacizumab and Axitinib
Number analyzed (Participants) | 70
months | 8.8 [8.1 to 10.2]

4. Secondary Outcome: Overall Survival (OS)
Description: Defined as the time from first treatment until death from any cause.
Time Frame: every 8 weeks until progression then every 3 months for up to 5 years.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FOLFOX/Bevacizumab and Axitinib
Number analyzed (Participants) | 70
months | 24.2 [16.0 to 30.9]

5. Secondary Outcome: Frequency of Adverse Events as a Measure of Safety
Description: The frequency of adverse events (AEs) was analyzed in 2 groups of patients, those receiving FOLFOX/bevacizumab (N=70), and patients who received axitinib maintenance (N = 48). AEs were assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.0.
Time Frame: Every 4 weeks plus 30 days during treatment and up to 5 years thereafter.
Measure: Number; unit: participants
Groups:
- FOLFOX/Bevacizumab: All patients who received at least one dose of FOLFOX/bevacizumab
- Axitinib: All patients who received at least one dose of axitinib
Arm/Group | FOLFOX/Bevacizumab | Axitinib
Number analyzed (Participants) | 70 | 49
participants
  Fatigue | 40 | 24
  Nausea | 37 | 15
  Diarrhea | 34 | 16
  Peripheral neuropathy | 34 | 16
  Neutropenia | 25 | 0
  Thrombocytopenia | 22 | 8
  Leukopenia | 21 | 7
  Anorexia | 19 | 14
  Mucositis | 18 | 5
  Proteinuria | 16 | 12
  Anemia | 16 | 7
  Constipation | 15 | 0
  Pain | 14 | 11
  Vomiting | 14 | 0
  Hypertension | 11 | 22
  Headache | 9 | 7
  Myalgia | 8 | 10
  Dizziness | 8 | 0
  Skin changes | 7 | 0
  Arthralgia | 7 | 6
  Hand-foot skin reaction | 0 | 7
  Dyspnea | 0 | 7
  Hoarseness | 0 | 7
  AST increased | 0 | 5

ADVERSE EVENTS:
Time Frame: Up to 3 years
Description: Safety population included all patients who received at least one dose of any study drug.
Arm/Group | FOLFOX/Bevacizumab and Axitinib
Serious Adverse Events (participants affected / at risk) | 13/70
Other Adverse Events (participants affected / at risk) | 70/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLFOX/Bevacizumab and Axitinib (N=70)
Chest pain (General disorders) | 2 (2) — There were two treatment-related deaths on study, due to reversible posterior leukoencephalopathy syndrome (RPLS) and febrile neutropenia/thrombocytopenia
Clostridium difficile colitis (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (2)
Intestinal obstruction (Gastrointestinal disorders) | 1 (2)
Tachycardia (Cardiac disorders) | 1 (2)
Accelerated hypertension (Vascular disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Embolism (Vascular disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Systemic candida (Infections and infestations) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FOLFOX/Bevacizumab and Axitinib (N=70)
Abdominal Pain (Gastrointestinal disorders) | 9
Alanine Aminotransferase Increased (Investigations) | 5
Alkaline Phosphatase Increased (Investigations) | 5
Allergic Reaction (Immune system disorders) | 6
Alopecia (Skin and subcutaneous tissue disorders) | 6
Anemia (Blood and lymphatic system disorders) | 18
Anorexia (Metabolism and nutrition disorders) | 24
Arthralgia (Musculoskeletal and connective tissue disorders) | 10
Aspartate Aminotransferase Increased (Investigations) | 5
Asthenia (General disorders) | 7
Chills (General disorders) | 4
Cold Intolerance (General disorders) | 4
Constipation (Gastrointestinal disorders) | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 7
Diarrhea (Gastrointestinal disorders) | 40
Dizziness (Nervous system disorders) | 9
Dysesthesia (Nervous system disorders) | 4
Dysgeusia (Nervous system disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Edema (General disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Fatigue (General disorders) | 48
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 5
Headache (Nervous system disorders) | 14
Hemorrhage (General disorders) | 4
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 8
Hypertension (Vascular disorders) | 27
Hypokalemia (Metabolism and nutrition disorders) | 7
Hypothyroidism (Endocrine disorders) | 4
Insomnia (Nervous system disorders) | 4
Leukopenia (Blood and lymphatic system disorders) | 25
Mucositis (Gastrointestinal disorders) | 18
Myalgia (Musculoskeletal and connective tissue disorders) | 13
Nausea (Gastrointestinal disorders) | 39
Neutropenia (Blood and lymphatic system disorders) | 26
Oral Pain (Gastrointestinal disorders) | 7
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 7
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 10
Paresthesia (Nervous system disorders) | 5
Peripheral Neuropathy (Nervous system disorders) | 41
Proteinuria (Renal and urinary disorders) | 20
Rash (Skin and subcutaneous tissue disorders) | 8
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 4
Skin Changes (Skin and subcutaneous tissue disorders) | 10
Sore Throat (Gastrointestinal disorders) | 5
Taste Alteration (Nervous system disorders) | 4
Temperature Intolerance (General disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 25
Vomiting (Gastrointestinal disorders) | 17
Weight Loss (Investigations) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.